CLINICAL TRIAL: NCT02561143
Title: To Evaluate the Effectiveness of Nutritional Counselling and "Improved Atta" Supplementation in Delaying Progression of Cachexia to Refractory Cachexia in Adult Cancer Patients in Indian Population
Brief Title: Effectiveness of Nutritional Counselling and "Improved Atta" Supplementation in Cachexic Adult Indian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Neha Kapoor, Research Scholar, University of Westminster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IEC/NP-339/08.10.2014
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Cachexia; Cancer
Keywords: cachexia; nutrition supplementation; IAtta; palliative care; quality of life
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Flour; Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will be given dietary supplement (Improved Atta: 100 g) daily along with nutritional counseling and physical activity counseling for six months.
  Interventions: Dietary Supplement: Improved Atta; Behavioral: Physical activity counseling; Other: Nutritional counseling
- Control group (Placebo Comparator): Patients in the control group will be given whole wheat flour (100 g) daily along with nutritional counseling and physical activity counseling for six months.
  Interventions: Dietary Supplement: Wheat flour; Behavioral: Physical activity counseling; Other: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Improved Atta — Improved Atta is a multi macro- micronutrient bread mix. Patients will be given 100 grams of Improved Atta (to make unleavened bread) everyday for consumption for six months.
  Arms: Intervention group
Dietary Supplement: Wheat flour — Whole wheat flour 100 grams (to make unleavened bread) will be given everyday for consumption for six months to the patients.
  Arms: Control group
Behavioral: Physical activity counseling — Depending on the physical status of the patients, low level of physical activity (walking and/or stairs), will be encouraged daily during counseling sessions.
Other: Nutritional counseling — Dietary counseling for 30 minutes will be imparted to all patients on every hospital visits by the nutritionist. Consumption of cereals, roots and tubers, vegetables, legumes, nuts, energy dense fruits, milk products (and eggs for non-vegetarians) will be encouraged in their daily diets.

SUMMARY:
Investigators are evaluating the nutritional role of IAtta supplementation along with nutritional counselling in delaying the progression of cachexia to refractory cachexia in adult cancer Indian patients. Patients will receive IAtta (100 g) or whole wheat flour (100 g) for daily consumption for 6 months. Dietary and physical activity counseling will be imparted every fortnight to patients.

Nutritional, biochemical, quality of life and anthropometric estimations will be assessed at baseline, after 3 months and at 6 months of intervention for all patients.

Investigators hypothesize that intake of nutrient rich bread mix IAtta (along with dietary and physical activity counselling) for six months will improve the health status and quality of life in free-living patients suffering from cancer cachexia.

DETAILED DESCRIPTION:
Patients will be randomly distributed into two groups i.e. control and intervention group. 75 patients will be allocated in intervention group and receive nutrient rich flour mix i.e. IAtta (100 g) along with dietary and physical activity counseling and 75 patients will be allocated in the control group who will receive whole wheat flour with dietary and physical activity counseling. Intervention group patients will collect 14 packets of 100 g of IAtta every fortnight during their clinician appointments while the control patients will collect 14 packets of 100 g of whole wheat flour at every clinician visit for 6 months.

Dietary counseling for 30 minutes will be imparted to all patients on each visit by the nutritionist. Depending on the physical status of the patients, low level of physical activity (walking and/or stairs), will be encouraged daily during counseling sessions.

Nutritional, biochemical, quality of life and anthropometric estimations would be assessed at baseline, after 3 months and at 6 months of intervention for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years and above.
* Diagnosed with cancer.
* Weight loss >5% from pre-treatment weight or BMI<20kg/m2.
* Hemoglobin level <12 g/dl.
* Energy intake < 1500 kcal/d (to be assessed on consultation)

Exclusion Criteria:

* Incapable to provide written consent.
* Patient diagnosed with refractory cachexia.
* Life expectancy < 3 months.
* Unresponsive to anti-cancer therapy.
* Patient is a pregnant woman or a nursing mother.
* Suffering from secondary illnesses.
* Gastrointestinal tract defects which affect nutrient absorption.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight at 6 months | Baseline, 3 months & 6 months
  Body weight in kilograms will be assessed using a Tanita segmental composition scale at baseline, mid-intervention (3 months) and at the end of intervention (6 months).

SECONDARY OUTCOMES:
Change in mid upper arm circumference (MUAC) at 6 months | Baseline, 3 months & 6 months
  MUAC in centimeters will be measured using a non-stretchable measuring tape at baseline, mid-intervention (3 months) and at the end of intervention (6 months).
Change in body fat percentage (BF%) at 6 months | Baseline, 3 months & 6 months
  Four site skin fold thickness (SFT) measurement (i.e. triceps, biceps, subscapular and suprailiac) by the help of scientific Harpenden Skinfold Caliper will be noted to the nearest 0.2mm reading, to calculate percentage body density. Body fat percentage will be calculated using body density value in Siri equation.
  SFT will be measured at baseline, mid-intervention (3 months) and end of intervention (6 months) to determine the BF%.
Indian Migrant study food frequency questionnaire (IMS-FFQ) | Baseline, 3 months & 6 months
  IMS-FFQ will be used to assess patient's daily energy (kcal), protein (g) and fat (g) intake at baseline, mid-intervention and end of intervention (6 months).
  Food frequency questionnaire is an accurate method to record the frequency of consumption of individual foods and can help provide information on patients' eating patterns. IMS-FFQ (Indian Migrant Study- Food Frequency Questionnaire) consists of 184 commonly consumed food items and is validated among the rural and urban Indian population.
Two day 24 hour dietary recall | Baseline, 3 months & 6 months
  Two day 24 hour dietary recall will be used to assess patient's daily energy (kcal), protein (g) and fat (g) intake at baseline, mid-intervention and end of intervention (6 months).
  24 hour dietary recall is an accurate method to understand patients' eating patterns.
Patient generated subjective global assessment (PGSGA) | Baseline, 3 months & 6 months
  PGSGA will be used to assess patient nutritional status (category: well nourished, malnourished & severely malnourished) at baseline, mid-intervention and end of intervention (6 months).
  PG-SGA is most effective and sensitive tool for assessing and evaluating cancer patients' nutritional status and validated on Indian cancer patients.
Indian Migrant Study Physical Activity Questionnaire (IMS-PAQ) | Baseline, 3 months & 6 months
  IMS-PAQ will assess patients' physical activity throughout the day. Investigators will asses physical activity at three time points during the study: baseline, at 3 months of intervention and at 6 months end of intervention. IMS-PAQ is a validated questionnaire on both Indian rural and urban population. Patients' will report every activity performed with the average amount of time spent for each activity in the questionnaire. Thereafter, investigators will calculate the average calories spent by every patient in the whole day.
Change in quality of life by EORTC-QLQ- C30 (Quality of life Questionnaire) at 6 months | Baseline, 3 months & 6 months
  EORTC-QLQ- C30 (European Organization for Research &Treatment of cancer) questionnaire will be used to analyse patients' quality of life at baseline, mid- intervention and at the end of intervention period. A score will be calculated for all the15 domains covered in the questionnaire of 30 questions.These domains will be analysed and compared for the outcome in the two groups.
Change in haemoglobin levels at 6 months | Baseline, 3 months & 6 months
  Haemoglobin levels (g/dl) will be monitored at baseline, at three months and at the end of intervention (6 months).
Change in serum albumin levels | Baseline, 3 months & 6 months
  Serum albumin (g%) levels will be monitored at baseline, at three months and at the end of intervention (6 months).
Change in C-reactive protein levels at 6 months | Baseline & 6 months
  C-reactive protein (mg/L) levels will be monitored at baseline and at the end of intervention (6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Neha Kapoor, PhD, Principal Investigator — University of Westminster; Ihab Tewfik, PhD, Study Director — University of Westminster
Locations (2):
- All India Institute of Medical Sciences, New Delhi, India
- University of Westminster, London, United Kingdom

REFERENCES:
- [Background] Kapoor N, Naufahu J, Tewfik S, Bhatnagar S, Garg R, Tewfik I. A public health nutrition intervention to delay the progression of cachexia to refractory cachexia in indian female cancer patients. Int. J. Food, Nutrition and Public Health. 2014;7:1-11.